CLINICAL TRIAL: NCT07340918
Title: Evaluation of the Association Between Incision and Suture Techniques Used in Abdominal Surgery and the Development of Incisional Hernia
Brief Title: Comparison of Small-bite Versus Conventional Midline Fascial Closure in Abdominal Surgeries
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Ilgaz Kayılıoğlu, Faculty Member, Muğla Sıtkı Koçman University
Other Study IDs: 06052021-10/I
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Incisional Hernia/Prevention and Control; Surgical Site Infection (SSI)
Keywords: incisional hernia; abdominal surgical procedures; wound closure techniques; postoperative complications
MeSH Terms: conditions — Incisional Hernia; Surgical Wound Infection; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional closure: This cohort includes patients who underwent midline abdominal fascial closure using the conventional closure technique as part of routine surgical practice. In this technique, the fascia was closed with continuous suturing using wider and deeper bites of the fascial edges and greater spacing between stitches compared with the small-bite approach. Closure was typically performed with a loop or single-strand absorbable monofilament suture and a larger needle, in accordance with traditional standards commonly applied in abdominal surgery.
  The choice of conventional closure was not randomized and reflected the operating surgeon's preference, intraoperative judgment, and case characteristics, such as incision length, wound conditions, and surgical urgency. This cohort therefore represents real-world clinical practice across a broad spectrum of elective and emergency abdominal procedures.
  No experimental intervention was assigned to this group. All other aspects of perioperative managemen
- Small-bite closure: This cohort includes patients who underwent midline abdominal fascial closure using the small-bite closure technique as part of routine surgical practice. In this technique, the fascia was closed with a continuous suture using small, closely spaced bites taken a short distance from the fascial edge, resulting in a higher suture-to-wound length ratio compared with conventional closure. An absorbable monofilament suture and a smaller needle were used, and stitches were placed at short intervals to achieve uniform tension distribution along the incision line.
  The selection of the small-bite technique was not randomized and depended on the operating surgeon's preference and intraoperative assessment. Prior to the initiation of the study, surgeons were familiar with and trained in the application of this technique, ensuring consistent execution within routine clinical practice. The cohort includes patients undergoing both elective and emergency abdominal procedures, reflecting everyday su

SUMMARY:
This study investigates how different incision and fascial closure (suture) techniques used in abdominal surgery are associated with the development of incisional hernia, a common long-term complication after laparotomy. Incisional hernia can cause pain, impaired quality of life, and may require additional surgery, making its prevention clinically important.

Adult patients undergoing midline abdominal surgery were followed prospectively. During surgery, detailed information about the incision and closure technique was recorded, including the type of fascial closure (small-bite versus conventional technique), incision length, suture length, and the suture-to-wound length ratio. Patient-related factors such as age, body mass index, comorbidities, and preoperative laboratory values were also collected. After surgery, patients were monitored for early wound complications, such as surgical site infection or wound dehiscence, and were followed for up to 12 months to assess whether an incisional hernia developed. Hernia diagnosis was based on clinical examination and ultrasonographic evaluation.

The main goal of the study is to identify which technical and patient-related factors are independently associated with the risk of incisional hernia. In particular, the study evaluates whether the small-bite fascial closure technique, which uses smaller and more closely spaced stitches, is associated with a lower risk of hernia formation and wound complications compared with conventional closure methods. Secondary objectives include assessing factors related to early postoperative wound complications and length of hospital stay.

By integrating surgical technique details with patient characteristics and postoperative outcomes, this study aims to improve understanding of modifiable risk factors for incisional hernia. The results may help surgeons choose closure techniques more effectively and improve postoperative outcomes for patients undergoing abdominal surgery.

DETAILED DESCRIPTION:
This study is designed as a prospective observational cohort investigation evaluating the relationship between abdominal incision characteristics, fascial closure (suture) techniques, and the subsequent development of incisional hernia following midline laparotomy. Incisional hernia represents one of the most frequent long-term complications after abdominal surgery and is associated with significant morbidity, impaired physical function, and the need for reoperation. Despite advances in surgical techniques, the relative contribution of technical factors and patient-related characteristics remains incompletely defined, particularly in heterogeneous populations that include both elective and emergency procedures.

Consecutive adult patients undergoing midline abdominal surgery were enrolled and followed longitudinally. The study does not involve randomization or protocol-driven assignment of surgical techniques; instead, closure methods were selected according to routine clinical practice and surgeon preference. Two commonly used fascial closure techniques were evaluated: the small-bite technique, characterized by closely spaced, shallow bites of the fascia, and the conventional technique, which uses wider and more widely spaced stitches. Intraoperative technical parameters were recorded in real time, including incision length, total suture length used for fascial closure, suture-to-wound length ratio, suture material, needle characteristics, and closure duration.

In addition to technical variables, comprehensive patient-related data were collected, including demographic characteristics, body mass index, comorbidity burden, surgical urgency (elective or emergency), wound classification, and relevant preoperative laboratory values reflecting nutritional and inflammatory status. Postoperatively, patients were monitored for early wound-related complications, such as surgical site infection, wound dehiscence, and evisceration, which were analyzed both individually and as a composite outcome.

Long-term follow-up was conducted using a standardized protocol. All participants were evaluated at 12 months after surgery for the presence of incisional hernia. Hernia assessment was based on structured clinical examination and confirmatory ultrasonographic imaging performed by study investigators. This approach was chosen to improve diagnostic accuracy and to capture both clinically apparent and subclinical hernias.

The primary outcome of the study is the occurrence of incisional hernia within 12 months of the index operation. Secondary outcomes include the development of early postoperative wound complications and duration of hospital stay. The analytical strategy focuses on identifying independent predictors of incisional hernia by integrating patient-related, intraoperative, and postoperative variables within multivariable statistical models. Particular emphasis is placed on evaluating whether specific closure techniques and quantitative measures of suturing, such as the suture-to-wound length ratio, are associated with reduced hernia risk after adjustment for potential confounders.

By systematically documenting real-world surgical practice and linking technical details to both short-term and long-term outcomes, this study aims to clarify modifiable factors that may reduce the incidence of incisional hernia. The findings are intended to support evidence-based decision-making in abdominal wall closure and to inform future strategies for improving surgical quality and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age) undergoing midline abdominal surgery
* Patients undergoing elective or emergency laparotomy
* Use of a midline abdominal incision with primary fascial closure
* Application of either small-bite or conventional fascial closure technique
* Availability of complete intraoperative data regarding incision and suture characteristics
* Provision of written informed consent
* Ability to participate in postoperative follow-up

Exclusion Criteria:

* Previous midline laparotomy or pre-existing incisional hernia
* Relaparotomy for indications other than incisional hernia
* Laparoscopic or minimally invasive procedures without midline fascial closure
* Presence of a pre-existing abdominal wall defect at the incision site
* Incomplete intraoperative data on closure technique or suture measurements
* Loss to follow-up or inability to complete 12-month postoperative assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients undergoing midline abdominal surgery at a tertiary referral general surgery center in Muğla. Participants were recruited consecutively from routine clinical practice and included individuals treated for a wide range of benign and malignant abdominal conditions. Both elective and emergency procedures were represented, reflecting the full spectrum of surgical activity at the study center.
  All operations were performed by experienced general surgeons using standardized perioperative care protocols. The population therefore represents a real-world cohort of patients treated in a high-volume surgical unit, encompassing variability in surgical urgency, wound conditions, and case complexity. Patients were followed prospectively within the same institution using a standardized postoperative and long-term follow-up program.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Incisional Hernia | 12 months
  The primary outcome measure was the occurrence of incisional hernia after midline abdominal surgery. Incisional hernia was defined as a postoperative defect of the abdominal wall at the site of the surgical incision, with or without a clinically visible or palpable bulge.
  All participants were followed prospectively using a standardized follow-up protocol. Assessment for incisional hernia was performed at 12 months after the index operation. Evaluation included a structured physical examination of the abdominal wall conducted by the study investigators. To increase diagnostic accuracy and to detect both clinically evident and subclinical hernias, all patients also underwent ultrasonographic examination of the incision site.
  The outcome was recorded as a binary variable (presence or absence of incisional hernia). Only hernias confirmed by clinical assessment and imaging were considered events. The time frame for outcome assessment was up to 12 months postoperatively.

SECONDARY OUTCOMES:
Early postoperative complications | 1 month
  Early postoperative complications were defined as wound-related adverse events occurring during the initial postoperative period following abdominal surgery. These complications included surgical site infection, wound dehiscence (partial separation of the wound), and fascial dehiscence or evisceration. Each complication was identified according to standard clinical criteria and documented prospectively during the hospital stay and early postoperative follow-up.
  Patients were routinely monitored through daily clinical examinations while hospitalized and during scheduled postoperative visits. When a wound-related complication was suspected, the diagnosis was confirmed based on clinical findings and, when necessary, additional investigations.
  For analysis, early postoperative complications were evaluated both as individual events and as a composite outcome representing the occurrence of any of the predefined wound complications. The outcome was recorded as a binary variable (presence o

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman Research and Training Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Plan Description
  Individual participant data (IPD) generated in this study include de-identified demographic information, perioperative clinical variables, intraoperative incision and closure characteristics, preoperative laboratory values, postoperative wound complications, and follow-up outcomes related to incisional hernia development. All shared data will be fully anonymized, with removal of direct and indirect identifiers, to protect participant confidentiality.
  IPD will not be made publicly available without restriction. Data may be shared with qualified researchers upon reasonable request, provided that approval is obtained from the relevant institutional ethics committee and that the proposed use is consistent with the original informed consent and ethical approvals of the study. Data sharing will be subject to a formal data use agreement defining the scope of use, data protection measures, and responsibilities of the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Tanriverdi E, Sahin S, Yazkan C, Dere O, Ozcan O, Kayilioglu I. Small-bite versus conventional midline fascial closure in abdominal surgery: a prospective observational cohort study. BMC Surg. 2026 Jan 24. doi: 10.1186/s12893-026-03530-x. Online ahead of print. PMID 41580707